CLINICAL TRIAL: NCT04888351
Title: Mastectomy and Breast Cancer : Follow-up of IBR's Rate and Study of Complications as Compared to Delayed Reconstructions Between 2016 and 2020 in Lyon
Brief Title: Immediate Breast Reconstruction's Increasing
Acronym: IBRI
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL21_0145
Record Dates: First submitted 2021-05-11; First posted 2021-05-17 (Actual); Last update posted 2021-05-17 (Actual); Status verified 2021-03

CONDITIONS: Breast Reconstruction; Breast Cancer
Keywords: Immediate Breast Reconstruction (IBR); Mastectomy; Breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Mastectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Mastectomies with IBR: Every women>18 years who underwent mastectomies followed by IBR (prothesis, latissimus dorsi flap, lipofeeling, isolated or combined) for breast cancer in Hôpital de la Croix-Rousse between January 2016 and January 2020
  Interventions: Other: Comparison of complications between mastectomies with IBR and mastectomies without IBR; Other: To analyze variations of number of patients eligibles to IBR
- Mastectomies without IBR: Every women>18 years who underwent mastectomies for breast cancer followed by delayed reconstructions (prothesis, latissimus dorsi flap, lipofeeling, isolated or combined) or no reconstructions between January 2016 and January 2020 in Hôpital de la Croix-Rousse
  Interventions: Other: Comparison of complications between mastectomies with IBR and mastectomies without IBR; Other: To analyze variations of number of patients eligibles to IBR

INTERVENTIONS:
Other: Comparison of complications between mastectomies with IBR and mastectomies without IBR — Precocious complications (less than 3 months after surgery) are classified with Clavien's classification : hematoma, seroma, stitches, antibiotics, transfusion.
  Tardive complications (after 3 months until 1 year) are more specifics : hematoma, seroma, tardive infections, asymmetry, removing of implant, breaking up of implant, skin necrosis, capsular contractures, implant loss, chronic pain.
Other: To analyze variations of number of patients eligibles to IBR — Including patients with differents classic risk factors : T3, T4, tobacco, diabetes, overweight and obesity, hypertension, age over 70, thoracic irradiation in the past

SUMMARY:
Mastectomy in breast cancer is still a way of treatment. Nowadays, the goal is to improve reconstruction's technicals. Immediate Breast Reconstruction (IBR) is one of them, largely used in United States but less in France. However, IGR (Insitut Gustave Roussey) in Paris just wrote a new protocole wich allows more IBR by including more patients.

This study aims to compare complications in 2 groups: mastectomies followed by IBR and mastectomies without IBR. The second goal will try to estimate the proportion of eligible's patients to IBR, and to analyse their surgicals and oncologicals risk factors

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years
* Breast cancer
* Mastectomy
* Hopital de la Croix-Rousse
* January 2016 and January 2020

Exclusion Criteria:

* Prophylactic mastectomy
* Male gender

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Female patients aged 18 or more, who have had a mastectomy for breast cancer in Croix-Rousse's hospital in Lyon, between 1st of January 2016 and 31st of December 2020
Sampling Method: Non-Probability Sample
Enrollment: 215 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-04-01 (Actual); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
Global complications's rates in 2 groups (percentage) | During first year after surgery
  Comparison of complications between mastectomies with IBR and mastectomies without IBR

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital de la Croix-Rousse, Lyon, France